CLINICAL TRIAL: NCT00356707
Title: Effect of Urban Form on Exercise and BMI in Black Women
Brief Title: Evaluating the Link Between Neighborhood Environments and Obesity Among African American Women
Status: Completed | Type: Observational
Sponsor: Boston University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1343; R01HL081399-01A1 (NIH); HL081399-01A1
Record Dates: First submitted 2006-07-25; First posted 2006-07-26 (Estimated); Last update posted 2012-03-28 (Estimated); Status verified 2012-03

CONDITIONS: Obesity
Keywords: Body Mass Index
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: This cohort comprises women from the Black Women's Health Study, a prospective study of African American women, who lived in the Los Angeles, New York, or Chicago metropolitan areas at the time of completion of the 1995, 1997, or 1999 questionnaires.

SUMMARY:
African American women have higher rates of obesity than women of any other racial or ethnic group in the United States. Obesity can have many causes, including genetic and environmental factors. This study will examine how neighborhood environments influence the occurrence of obesity among African American women.

DETAILED DESCRIPTION:
Obesity, which leads to higher rates of diabetes, cancer, and heart disease, is an increasingly important public health problem. In 2000, over 78% of African American women were overweight, and over 50% were obese. Several factors can contribute to obesity, including genetics, diet, and environmental factors. Individuals who live in an environment in which it is difficult to maintain an active lifestyle are more prone to obesity. The Black Women's Health Study (BWHS) is an extensive long-term study that is gathering data from women across the country to examine the occurrence of various diseases among African American women. Using BWHS study data and specific information on participants' neighborhoods, including street layout and the presence of sidewalks, this study will determine if neighborhood environments influence the prevalence of obesity among African American women.

This study will use already-collected data on physical activity and body mass index of BWHS study participants who live in New York, Los Angeles, and Chicago; there are no additional study visits specifically for this study. A transportation and urban planning expert will compile data regarding the pedestrian environment of neighborhoods in all three cities, including the nature and density of land use, proximity to parks, presence of sidewalks, speed and volume of traffic, and street structure. Census data regarding participants' socioeconomic status will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Participating in the BWHS study
* Residing in New York, Los Angeles, or Chicago

Ages: 21 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The Black Women's Health Study cohort comprises 59,000 African American women recruited mainly from subscribers to Essence magazine who returned the baseline 1995 survey.
Sampling Method: Non-Probability Sample
Enrollment: 23000 (Actual)
Dates: Start 2006-06; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Influence of neighborhood environments on obesity among African American women | Measured through the use of BWHS study data and neighborhood study data

CONTACTS AND LOCATIONS:
Overall Officials: Patricia F. Coogan, ScD, Principal Investigator — Boston University
Locations (1):
- Slone Epidemiology Center, Boston University, Boston, Massachusetts, United States